CLINICAL TRIAL: NCT06831461
Title: Proton Versus Photon Radiotherapy In Adults With Primary Brain Tumors Evaluating Functional Survival: A Phase 3 Randomized Controlled Trial (PRIDE)
Brief Title: Proton Versus Photon Radiotherapy in Adults With Primary Brain Tumors
Acronym: PRIDE
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Tata Memorial Centre (Other)
Responsible Party: Principal Investigator, Dr Archya Dasgupta, Associate Professor in Department of Radiation Oncology, Tata Memorial Centre
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 4617
Record Dates: First submitted 2025-02-12; First posted 2025-02-18 (Actual); Last update posted 2025-09-16 (Actual); Status verified 2025-09

CONDITIONS: Primary Brain Tumors; Diffuse Glioma; Meningioma; Pituitary Adenoma; Low Grade CNS Tumors
Keywords: Proton Beam Therapy; Photon Radiotherapy; Brain Tumors; Neurocognition; Survival
MeSH Terms: conditions — Brain Neoplasms; Meningioma; Pituitary Neoplasms | interventions — Proton Therapy

STUDY DESIGN:
Intervention Model Description: Prospective, open-label, superiority, 2-arm, randomized controlled trial, phase 3 study.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Photon therapy (standard arm) (Other): Patients in the standard arm will undergo focal cranial radiotherapy using photons (X-rays) with image guidance using IMRT, VMAT, or helical intensity-modulated techniques.
  Interventions: Radiation: Photon Radiotherapy
- Proton beam therapy (experimental arm) (Experimental): The patients in the experimental arm will undergo focal radiotherapy to an equivalent dose using proton beam therapy.
  Interventions: Radiation: Proton Beam Therapy

INTERVENTIONS:
Radiation: Proton Beam Therapy — Patients randomized to the experimental arm will be treated with proton beam therapy.
  Arms: Proton beam therapy (experimental arm)
Radiation: Photon Radiotherapy — Patients randomized to standard arm will be treated with photon therapy.
  Arms: Photon therapy (standard arm)

SUMMARY:
This study will be done in adults with brain tumors having good prognosis requiring treatment with radiotherapy. The current practice for brain radiotherapy involves treatment using X rays (photon radiotherapy). Proton beam therapy is a more advanced form of delivering radiation, which allows the reduction of the dose of radiation to the parts of the brain surrounding the tumor. After treatment with photon radiotherapy, certain late effects of radiation, like memory decline, hormonal deficits, hearing loss, and worsening of neurological function, can occur in some patients. From the evaluation of dose profiling, proton beam therapy has the potential to reduce the possibility of side effects by reducing the dose to critical organs. However, there is no clinical data to demonstrate whether the theoretical dose reduction translates to a clinically meaningful benefit. In the proposed study, 156 patients will be randomly allocated to either proton or photon radiotherapy in 1: 1 ratio. The primary objective of the study is to explore whether proton therapy improves functional survival, which is life expectancy without recurrence, death, or complications from radiotherapy.

DETAILED DESCRIPTION:
Patients aged 18 to 70 years who are planned for focal cranial radiotherapy for primary CNS tumors meeting eligibility criteria will be considered for the study. Indications for radiation will be as per standard institutional practice, primarily decided by histology, tumor grade, molecular features (as appropriate for selected histologies), type of tumor resection, and extent of disease. Patients with an expected life expectancy of more than 5 years, as per published literature and institutional data, will be considered eligible for the study. This will include but is not limited to the diagnosis of low-grade glial/ glioneural tumors, IDH-mutant grade 2/3 gliomas (astrocytoma and oligodendroglioma), ependymoma, meningioma, pituitary tumor, craniopharyngioma, schwannoma. In some instances, which are treated based on a radiological diagnosis (without needing a histopathological diagnosis), like schwannoma, meningioma will be eligible for the study. After discussion with patients and caregivers, consent forms will be served and accrued in the study once a signed consent form is obtained. Randomization will be done in a 1:1 ratio by the statistician via computerized software using a permuted block design accounting for the stratification factors mentioned earlier.

Patients in the standard arm will undergo focal cranial radiotherapy using photons (X-rays) with image guidance using IMRT, VMAT, or helical intensity-modulated techniques. The patients in the experimental arm will undergo focal radiotherapy to an equivalent dose using protons with pencil beam scanning or volumetric modulated proton arc therapy. The radiation dose and volumes will be guided by tumor type and molecular features without any influence from the current study on radiation protocols. Baseline workup investigations for diagnosis and treatment plan will be undertaken per standard practice, including histopathological evaluation, molecular evaluation, blood analysis, and imaging with magnetic resonance imaging (MRI) brain tumor protocol. Patients will be simulated in a supine position and immobilized using head-neck thermoplastic masks fitted to a Universal Base Plate according to the institutional protocol and the arm randomized (as appropriate for proton or photon therapy). Radiation planning non-contrast computed tomography (NCCT) scan will be acquired from the top of the vertex to the clavicle with a slice thickness of 1.25-2.5 mm. Planning MRI of the brain will be done per institutional practice, including 3D sequences of T1-contrast, 3D T2-weighted propellor, 3D T2-FLAIR sequences, and additional sequences like FIESTA or CISS as indicated (for skull base targets) is needed within 4 weeks from starting radiation. Planning PET scans will be done in patients with tumor diagnosis of meningioma, schwannoma, and pituitary tumors as clinically indicated.

The contouring of target volumes will be done by the radiation oncologists using registrations of appropriate planning imaging to delineate gross tumor volume (GTV), clinical target volume (CTV), and planning target volumes (PTV) as applicable for the tumor type without any influence of the study arm. Organs at risk (OAR) like the hippocampus, temporal lobes, amygdala, brainstem, optic nerves and optic chiasm, pituitary gland, cochlea, oral cavity, eye, lens, etc., will be contoured for the plan as per institutional practice.Dose prescriptions will be done as per standard practice. Typically, the target volume dose prescriptions currently for the common histologies likely to be included in the study are as follows: diffuse gliomas (55.8 Gy-59.4 Gy using 1.8 Gy per fraction depending upon subtype i.e., oligodendroglioma vs. astrocytoma); ependymoma (59.4 Gy using 1.8 Gy per fraction), meningioma (54 Gy to 60 Gy using 1.8/2 Gy per fraction depending upon grade, location, molecular features); craniopharyngioma, schwannoma (54 Gy in 30 fractions); circumscribed glioma, low-grade glioma (50 Gy to 54 Gy in 1.67/ 1.8 Gy depending upon location); pituitary tumors (45 Gy in 25 fractions).To avoid any potential bias from the study arm, the dose fractionation needs to be defined before randomization, which also serves as a stratification factor. The OAR tolerance will be used as per standard practice and existing literature. The radiation plan will be made in the Treatment Planning System (TPS) by designated medical physicists and reviewed by the responsible radiation oncologist. Given the diverse location of the target volumes for patients accrued in the study, no predefined dose-volume constraints are mandated. However, the principle of low as reasonably achievable (ALARA) will be followed by practicing reasonable dose-volume constraints as per current literature and institutional practice. As a part of quality assurance, the radiation target volume and plan will be individually reviewed in the radiation-planning review meeting, comprising radiation oncologists, medical physicists, neuroradiologists, and radiation therapy technologists. Treatment will be delivered on photon or proton facilities equipped with image guidance platforms. All patients will be reviewed on a weekly basis by radiation oncologists to monitor for acute radiation-related toxicities. Interval imaging and adaptive planning will be done as per standard practice in both study arms without any influence from the study participation. Chemotherapy (concurrent or adjuvant) will be given as indicated (IDH-mutant glioma).

After completion of radiotherapy, patients will undergo scheduled regular clinical and radiological follow-ups as per standard practice without any influence from the study. The first imaging after radiation for IDH-mutant gliomas is done 1-month post-radiotherapy, before starting adjuvant chemotherapy, and after that during adjuvant chemotherapy and at the conclusion. Otherwise, for high-grade tumors (not planned for adjuvant chemotherapy) treated with radiation, the first imaging is done 1-2 months, while for low-grade and benign tumors, it is done 2-3 months after completion of radiotherapy. As per standard practice, after completing all scheduled treatments (including chemotherapy), patients will undergo scheduled clinical evaluation every 3-6 months for the initial 2 years and every 6 months after that. Institutional protocols include surveillance imaging every 6-12 months for high-grade tumors and every 12 months for low-grade tumors or as per clinical indication (during new symptoms), which will be applicable to the current study. Patients are not required to have any additional visits for study-related purposes. Any disease recurrence or complications arising from treatments will be treated as per standard practice and discussion in the joint neuro-oncology clinic as required.

Functional assessments:

The time points for functional assessment will be as per standard institutional, which is discussed below. Neurocognitive evaluation using age-appropriate tests by psychologists will include the Wechsler Adult Intelligence Scale test, which provides the Full-Scale Intelligence Quotient (FSIQ) and other subdomains as the Verbal Quotient (VQ), Performance Quotient (PQ). Neurocognitive assessment will be done before starting radiotherapy (baseline), post-radiotherapy 6 months, 1 year, and annually after that. To evaluate the endocrine function, the pituitary profile will be tested, which includes thyroid-stimulating hormone, free T4, T3, insulin-like growth factor (IGF)-1, growth hormone (GH), estrogen, testosterone, follicle-stimulating hormone (FSH), luteinizing hormone (LH), adrenocorticotropic hormone (ACTH), cortisol, and prolactin levels will be assessed.

The auditory function will be tested using pure tone audiometry. Endocrinal and auditory assessments will be done before starting radiation and annually after that. Patient-reported outcomes will be recorded using the EORTC QLQ core (C-30) and brain (BN-20) modules for quality-of-life assessment before starting radiation, once during mid-radiotherapy (3rd to 4th week), at conclusion, 1-3 months after completion (during 1st follow-up visit after radiotherapy), 6 months, 1 year after completion, and annually after that. The sleep and dream will be assessed the PSQI and MADRE questionnaires, respectively. The timepoints of assessment will be similar to QOL assessments.

All pre-radiation (baseline) investigations are required to be done within 1 month before the start of the radiotherapy.

Oncological and toxicity assessments: The assessment of disease status and radiation-induced toxicity in the form of radionecrosis will be done by serial clinical and imaging surveillance, as outlined earlier. In equivocal cases of radionecrosis, additional imaging with amino acid PET will be done and discussed in the multidisciplinary joint neuro-oncology meeting. Disease progression will be defined by the response assessment in neuro-oncology (RANO) 2.0 criteria.

ELIGIBILITY:
Inclusion Criteria:

* Primary brain tumors
* Age at irradiation: 18 to 70 years
* Karnofsky Performance Status ≥ 60
* Diagnosis (histopathological/ radiological) of primary brain tumor with an expected survival of >5 years (e.g., grade 2-3 diffuse glioma, low-grade glial/ glioneuronal tumors, ependymoma, meningioma, pituitary tumors, schwannoma, craniopharyngioma, etc.)
* Planned for focal cranial radiotherapy
* Informed consent taken

Exclusion Criteria:

* Re-irradiation
* Palliative radiotherapy
* Multifocal or multicentric disease
* Planned for whole brain irradiation or craniospinal irradiation
* Planned for hypo-fractionated or stereotactic radiotherapy

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 156 (Estimated)
Dates: Start 2025-07-01 (Actual); Primary Completion 2032-12-31 (Estimated); Study Completion 2032-12-31 (Estimated)

PRIMARY OUTCOMES:
5-year functional survival | 7 years
  Functional survival will be calculated using Kaplan Meier method from the date of randomization as the primary outcome for the study. Any of the following will be considered as an event for the assessment of functional survival.
  1. Cognitive decline: A drop of 10% from baseline in the FSIQ or any sub-domains of the neurocognition test.
  2. CTCAE v.5 gr ≥2 ototoxicity: Threshold shift of >25 dB averaged at 2 or more contiguous test frequencies in at least one ear (on a 1, 2,3,4,6 and 8kHz audiogram) or decrease in hearing to profound bilateral loss.
  3. Endocrinal dysfunction: Significant decline in one or multiple pituitary axes and/or starting/increasing dose of hormone supplements.
  4. Neurological impairment: A decrease in the NPS by 2 points or KPS by atleast 30 points from pre-radiation status.
  5. CTCAE gr ≥3 radio-necrosis
  6. Disease progression
  7. Death

SECONDARY OUTCOMES:
Overall Survival | 7 years
  Overall survival will be calculated using Kaplan Meier method with death from any cause considered as an event.
Progression free survival | 7 years
  Progression free survival will be calculated using Kaplan Meier method with disease progression considered as an event.
Acute radiation toxicity | 7 years
  The cumulative incidence of acute radiation toxicity (upto 90 days from completion of radiotherapy) will be compared between the two study arms using Chi-square test
Quality of life core questionnaire | 7 years
  The European Organization for Research and Treatment of Cancer (EORTC) quality of life (QOL) core questionnaire (C30) will be used. The summary scores will be calculated from the raw scores as per the manual, ranging from 0 to 100, with higher scores representing better outcomes. The global score and scores of subdomains will be calculated during follow-up and compared with baseline.
Quality of life brain cancer module | 7 years
  The European Organization for Research and Treatment of Cancer (EORTC) brain module (BN20) questionnaire will be used. The summary scores will be calculated from the raw scores as per the manual, ranging from 0 to 100, with higher scores representing better outcomes. The global score and scores of subdomains will be calculated during follow-up and compared with baseline.
Cost-benefit analysis | 7 years
  Cumulative cost of radiation treatment and cost of management of acute or delayed side effects between the two groups will be compared using proportions of expenditure.

CONTACTS AND LOCATIONS:
Locations (1):
- Tata Memorial Centre, Mumbai, India

IPD SHARING:
Plan to Share IPD: No
IPD will be shared upon reasonable request to the principal investigator following institutional ethics committee guidelines.